CLINICAL TRIAL: NCT01209195
Title: A Phase 1, Pharmacologic and Pharmacodynamic Study of MM-121 in Combination With Paclitaxel in Patients With Advanced Gynecologic and Breast Cancers
Brief Title: A Study of MM-121 in Combination With Paclitaxel in Patients With Advanced Gynecologic and Breast Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-121-04-01-04
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Results first posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Locally Advanced/Metastatic or Recurrent Ovarian Cancer, Fallopian Tube Cancer,; Primary Peritoneal Cancer or Endometrial Cancer; Locally Advanced/Metastatic Her2 Non Overexpressing Breast Cancer
Keywords: Ovarian cancer; HER-2 negative breast cancer; Breast cancer; Fallopian tube cancer
MeSH Terms: conditions — Neoplasm Metastasis; Ovarian Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms; Breast Neoplasms | interventions — seribantumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MM-121 + Paclitaxel (Experimental): Escalating doses of MM-121 given IV QW in combination with paclitaxel at standard dose of 80 mg/m2 IV QW
  Interventions: Drug: MM-121; Drug: Paclitaxel

INTERVENTIONS:
Drug: MM-121 — increasing doses of MM-121 IV QW
  Other Names: Seribantumab, SAR256212
Drug: Paclitaxel — Paclitaxel - 80 mg/m2 IV QW
  Other Names: Taxol

SUMMARY:
This study was a Phase 1 and pharmacologic open-labeled dose-escalation trial of MM-121 in combination with paclitaxel using a "3+3" design.

DETAILED DESCRIPTION:
Successive cohorts of three or more patients were treated at escalating doses until a maximum tolerated dose/recommended phase 1 dose was identified. Once the maximum tolerated dose was identified, an Expansion Cohort was enrolled at that dose to further characterize safety and to explore pharmacodynamic endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Cytological or histological confirmation of locally advanced/metastatic or recurrent epithelial ovarian cancer, fallopian tube cancer, primary peritoneal cancer or endometrial cancer; OR, cytological or histological confirmation of locally advanced /metastatic Her2 non-overexpressing breast cancer
* Eighteen years of age or above
* Candidates for chemotherapy
* Able to understand and sign an informed consent (or have a legal representative who is able to do so)
* Measurable disease according to RECIST v1.1
* ECOG Performance Score (PS) of ≤ 2
* Willing to abstain from sexual intercourse or to use an effective form of contraception during the study and for 90 days following the last dose of MM-121

Exclusion Criteria:

* Prior radiation therapy to >25% of bone marrow-bearing areas
* Evidence of any other active malignancy
* Active infection or fever> 38.5°C during screening visits or on the first scheduled day of dosing
* Symptomatic CNS disease
* Known hypersensitivity to any of the components of MM-121 or who have had hypersensitivity reactions to fully human monoclonal antibodies
* Received treatment, within 30 days prior to the first scheduled day of dosing, with any investigational agents that have not received regulatory approval for any indication or disease state
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-10; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akos Czibere, MD, PhD, Study Director — Merrimack Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Cancer Care Associates of Fresno, Fresno, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Dose Escalation: Cohort 1: MM-121 - 20 mg/kg loading dose followed by 12 mg/kg weekly IV Paclitaxel - 80mg/m2 weekly IV
- Part 1: Dose Escalation: Cohort 2; Part 2: Expansion Cohort 1: MM-121 - 40 mg/kg loading dose followed by 20 mg/kg weekly IV
  Paclitaxel - 80mg/m2 weekly IV
- Part 2: Expansion Cohort 2: MM-121 20 mg/kg IV loading dose followed by 12 mg/kg IV QW maintenance dose
  Paclitaxel: 80 mg/m2 weekly IV
- Part 2: Cohort 3: MM-121 40mg/kg IV QOW
  Paclitaxel: 80 mg/m2 weekly IV
- Part 2: Cohort 4: MM-121 - 40 mg/kg loading dose followed by 20 mg/kg weekly IV for 3 weeks, followed by one week of rest
  Paclitaxel - 80mg/m2 weekly IV for 3 weeks, followed by one week of rest
Period: Overall Study
Arm/Group | Part 1: Dose Escalation: Cohort 1 | Part 1: Dose Escalation: Cohort 2 | Part 2: Expansion Cohort 1 | Part 2: Expansion Cohort 2 | Part 2: Cohort 3 | Part 2: Cohort 4
Started | 7 | 3 | 6 | 6 | 6 | 13
Completed | 7 | 3 | 6 | 6 | 6 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MM-121 + Paclitaxel: Dose Escalation: MM-121 plus Paclitaxel: Cohort 1:
  MM-121 - 20 mg/kg loading dose followed by 12 mg/kg weekly IV Paclitaxel - 80mg/m2 weekly IV
  Cohort 2:
  MM-121 - 40 mg/kg loading dose followed by 20 mg/kg weekly IV Paclitaxel - 80mg/m2 weekly IV
  Intermediate doses between cohorts 1 and 2 may also be considered.
- MM-121 + Paclitaxel: Expansion Cohort: MM-121 - 40 mg/kg loading dose followed by 20 mg/kg weekly IV Paclitaxel - 80mg/m2 weekly IV
- Total: Total of all reporting groups
Arm/Group | MM-121 + Paclitaxel: Dose Escalation | MM-121 + Paclitaxel: Expansion Cohort | Total
Number analyzed (Participants) | 10 | 31 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (9.62) | 55.5 (10.43) | 56.45 (10.025)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 31 | 41
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 10 | 11
  Not Hispanic or Latino | 9 | 21 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 10 | 22 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 5 | 5
Region of Enrollment [Number; unit: participants]
  United States | 10 | 31 | 41

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation: To Evaluate the Safety and Tolerability of Escalating Doses of the MM-121 Plus Paclitaxel Combination Via Reporting of Dose-limiting Toxicity (DLT)
Description: To establish the safety of escalating doses of MM-121 in combination with paclitaxel in order to determine the recommended phase 2 dose. Dose-escalation conducted using standard 3+3 model to determine maximum tolerated dose. Reports of Dose-Limiting Toxicities (DLTs) were assessed to determine the MTD.
Time Frame: From date of first dose to 30 days after termination, the longest 163 weeks
Measure: Number; unit: participants reporting DLTs
Arm/Group | Part 1: Dose Escalation: Cohort 1 | Part 1: Dose Escalation: Cohort 2 | Part 2: Expansion Cohort 1 | Part 2: Expansion Cohort 2 | Part 2: Cohort 3 | Part 2: Cohort 4
Number analyzed (Participants) | 7 | 3 | 6 | 6 | 6 | 13
participants reporting DLTs | 0 | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: To Determine the Maximum Tolerated Dose (MTD) of MM-121 in Combination With Paclitaxel: MM-121 Dose Level
Description: Using a 3+3 dose escalation model, the maximum tolerated dose of each combination was determined by assessing dose-limiting toxicities in each cohort.
  Part 1 Cohort 1: MM-121: 20 mg/kg loading dose followed by 12 mg/kg QW IV )20/12) + Paclitaxel: 80mg/m2 IV QW Part 1 Cohort 2: MM-121: 40 mg/kg loading dose followed by 20 mg/kg QW IV (40/20) + Paclitaxel: 80mg/m2 QW IV Part 2 Cohort 1: MM-121: 40/20 mg/kg IV + Paclitaxel: 80mg/m2 QW IV Part 2 Cohort 2: MM-121 20 /12 mg/kg IV QW + Paclitaxel: 80 mg/m2 QW IV Part 2 Cohort 3: MM-121 40mg/kg IV QOW + Paclitaxel: 80 mg/m2 QW IV Part 2 Cohort 4: MM-121 - 40 mg/kg loading dose followed by 20 mg/kg weekly IV for 3 weeks, followed by one week of rest + Paclitaxel: 80mg/m2 weekly IV for 3 weeks, followed by one week of rest
Time Frame: From date of first dose to 30 days after termination, the longest 163 weeks
Population: NOTE: MTD of paclitaxel when administered with MM-121 provided in separate endpoint entry
Measure: Number; unit: mg/kg
Groups:
- Part 1: Dose Escalation: Escalating doses of MM-121 and paclitaxel
- Part 2: Expansion Cohorts: Additional exploratory doses of MM-121 and paclitaxel
Arm/Group | Part 1: Dose Escalation | Part 2: Expansion Cohorts
Number analyzed (Participants) | 10 | 31
mg/kg
  one-time loading dose | 40 | 40
  maintenance dose | 20 | 20

3. Primary Outcome: To Determine the Maximum Tolerated Dose (MTD) of MM-121 in Combination With Paclitaxel: Paclitaxel Dose Level
Description: as for outcome 2
Time Frame: From date of first dose to 30 days after termination, the longest 163 weeks
Population: note: MTD of MM-121 when administered in combination with paclitaxel provided in separate endpoint entry
Measure: Number; unit: mg/m2
Arm/Group | Part 1: Dose Escalation | Part 2: Expansion Cohorts
Number analyzed (Participants) | 10 | 31
mg/m2 | 80 | 80

4. Secondary Outcome: To Characterize the Efficacy of the Combination of MM-121 and Paclitaxel Using Objective Response Rate
Description: To determine the number of patients reporting an objective response using RECIST v 1.1 where a Partial Response (PR) is defined as >20% decrease in tumor burden from baseline and a Complete Response (CR) is defined as complete disappearance from tumor burden from baseline. Objective Response is presented as the total # patients with PR or CR.
Time Frame: patients were assessed for response during their time on study, the longest of which was 163 weeks
Measure: Number; unit: participants with objective response
Arm/Group | Part 1: Dose Escalation: Cohort 1 | Part 1: Dose Escalation: Cohort 2 | Part 2: Expansion Cohort 1 | Part 2: Expansion Cohort 2 | Part 2: Cohort 3 | Part 2: Cohort 4
Number analyzed (Participants) | 7 | 3 | 6 | 6 | 6 | 13
participants with objective response | 1 | 2 | 3 | 3 | 3 | 2

5. Secondary Outcome: To Determine the Pharmacokinetics (PK) of MM-121 When Administered in Combination With Paclitaxel
Description: Pharmacokinetic (PK) evaluation was performed on plasma samples obtained weekly for the first cycle of the study and then on day 1 of each additional cycle to assess pre-treatment trough concentrations of MM-121. Non-compartmental analysis (NCA) was performed to calculate standard PK parameters, including the maximum observed concentration (Cmax). Serum levels of MM-121 were measured at a central lab using an enzyme-linked immunosorbent assay (ELISA). Data is presented per dose level of MM-121 (20/12 mg/kg weekly, 40/20 mg/kg weekly, 40 mg/kg Q2W, or 40/20 mg/kg QW x 7 plus a rest week).
Time Frame: Collections taken at for all patients at Cycle 1, Week 1 (pre-treatment/pre-infusion, at the end of the infusion, and 2.5, 4, 6 and 24 hours after starting the infusion of MM-121) and pre-treatment at Cycle 1, Week 3 and Cycle 2, Week 1
Population: All patients. Data presented per dose level of MM-121 and not per cohort. The same dose was used in multiple cohorts, and those data were combined.
  NOTE: two patients are not included in the analysis due to incorrectly collected or processed samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Groups:
- MM-121 + Paclitaxel: 20/12 mg/kg: MM-121: 20 mg/kg loading dose followed by 12 mg/kg weekly maintenance dose Paclitaxel: 80 mg/m2
- MM-121 + Paclitaxel: 40/20 mg/kg: MM-121: 40 mg/kg loading dose followed by 20 mg/kg weekly maintenance dose Paclitaxel: 80 mg/m2
- MM-121 + Paclitaxel: 40 mg/kg Q2W: MM-121: 40 mg/kg Q2W Paclitaxel: 80 mg/m2
- MM-121 + Paclitaxel: 40/20 mg/kg + Rest Week: MM-121: 40 mg/kg loading dose followed by seven 20mg/kg weekly doses and a rest week. This administration schedule spans two cycles and repeats for each subsequent 2-cycle unit.
  Paclitaxel: 80 mg/m2
Arm/Group | MM-121 + Paclitaxel: 20/12 mg/kg | MM-121 + Paclitaxel: 40/20 mg/kg | MM-121 + Paclitaxel: 40 mg/kg Q2W | MM-121 + Paclitaxel: 40/20 mg/kg + Rest Week
Number analyzed (Participants) | 12 | 9 | 6 | 12
ug/mL | 445.7 (39.6) | 903.5 (31.5) | 1081.1 (73.1) | 1134.5 (18.6)

6. Secondary Outcome: Pharmacokinetic Parameters (AUClast)
Description: Pharmacokinetic (PK) evaluation was performed on plasma samples obtained weekly for the first cycle of the study and then on day 1 of each additional cycle to assess pre-treatment trough concentrations of MM-121. Non-compartmental analysis (NCA) was performed to calculate standard PK parameters, including the maximum observed concentration (Cmax). Serum levels of MM-121 were measured at a central lab using an enzyme-linked immunosorbent assay (ELISA). Data is presented per dose level of MM-121 (20/12 mg/kg weekly, 40/20 mg/kg weekly, 40 mg/kg Q2W, or 40/20 mg/kg QW x 7 plus a rest week).
  Immunogenicity data is not available.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr* ug/mL
Arm/Group | MM-121 + Paclitaxel: 20/12 mg/kg | MM-121 + Paclitaxel: 40/20 mg/kg | MM-121 + Paclitaxel: 40 mg/kg Q2W | MM-121 + Paclitaxel: 40/20 mg/kg + Rest Week
Number analyzed (Participants) | 12 | 9 | 6 | 12
hr* ug/mL | 39252.9 (40.3) | 77137.6 (31.1) | 102263.1 (35.6) | 96043.0 (25.9)

7. Secondary Outcome: Immunogenicity
Description: Samples were collected to determine the presence of an immunologic reaction to MM-121 (i.e. human anti-human antibodies).
Time Frame: Samples were collected for all patients pre-dose on all cycles for duration of treatment, the longest of which was 163 weeks, and a collection was made post-infusion in any case of infusion reaction
Measure: Number
Arm/Group | Part 1: Dose Escalation: Cohort 1 | Part 1: Dose Escalation: Cohort 2 | Part 2: Expansion Cohort 1 | Part 2: Expansion Cohort 2 | Part 2: Cohort 3 | Part 2: Cohort 4
Number analyzed (Participants) | 7 | 3 | 6 | 6 | 6 | 13
Value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value

ADVERSE EVENTS:
Time Frame: AEs were collected from a patient's first dose until 30 days after treatment termination. SAEs were collected from time of informed consent until 30 days after termination. If related, events could be reported at any time after termination.
Description: All related AEs ongoing at the time of treatment discontinuation were followed until resolution. Investigators were to report any AEs/SAEs assumed to be related any time, even if occurring more than 30 days after last dose. Though different for each patient, on average, patients could be followed for related AEs/SAEs for ~1 year after termination
Groups:
- MM-121 + Paclitaxel: Dose Escalation: Cohort 1:
  MM-121 - 20 mg/kg loading dose followed by 12 mg/kg weekly IV Paclitaxel - 80mg/m2 weekly IV
  Cohort 2:
  MM-121 - 40 mg/kg loading dose followed by 20 mg/kg weekly IV Paclitaxel - 80mg/m2 weekly IV
- MM-121 + Paclitaxel: Expansion Cohort: Cohort 1:
  MM-121 - 40 mg/kg loading dose followed by 20 mg/kg weekly IV Paclitaxel - 80mg/m2 weekly IV
  Cohort 2:
  MM-121 20 mg/kg IV loading dose x followed by 12 mg/kg IV QW maintenance dose Paclitaxel: 80 mg/m2 weekly IV
  Cohort 3:
  MM-121 40mg/kg IV QOW Paclitaxel: 80 mg/m2 weekly IV
  Cohort 4:
  MM-121 - 40 mg/kg loading dose followed by 20 mg/kg weekly IV for 3 weeks, followed by one week of rest Paclitaxel - 80mg/m2 weekly IV for 3 weeks, followed by one week of rest
Arm/Group | MM-121 + Paclitaxel: Dose Escalation | MM-121 + Paclitaxel: Expansion Cohort
Serious Adverse Events (participants affected / at risk) | 4/10 | 12/31
Other Adverse Events (participants affected / at risk) | 10/10 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MM-121 + Paclitaxel: Dose Escalation (N=10) | MM-121 + Paclitaxel: Expansion Cohort (N=31)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 | 0 — Any Relationship
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 — Any Relationship
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0 — Any Relationship
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 — Any Relationship
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 — Any Relationship
GASTRITIS (Gastrointestinal disorders) | 0 | 1 — Any Relationship
PEPTIC ULCER (Gastrointestinal disorders) | 0 | 1 — Any Relationship
DEATH (General disorders) | 1 | 0 — Any Relationship
DISEASE PROGRESSION (General disorders) | 0 | 3 — Any Relationship
FATIGUE (General disorders) | 0 | 2 — Any Relationship
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 — Any Relationship
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 — Any Relationship
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Any Relationship
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 — Any Relationship
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 2 — Any Relationship
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Any Relationship
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 1 | 0 — Any Relationship
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 2 — Any Relationship
HEPATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1 — Any Relationship
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1 — Any Relationship
SEPSIS (Infections and infestations) | 0 | 1 — Any Relationship
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Any Relationship
THROMBOSIS (Vascular disorders) | 0 | 1 — Any Relationship
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MM-121 + Paclitaxel: Dose Escalation (N=10) | MM-121 + Paclitaxel: Expansion Cohort (N=31)
ABDOMINAL PAIN (Gastrointestinal disorders) | 9 | 7 — Any Relationship
DIARRHOEA (Gastrointestinal disorders) | 5 | 18 — Any Relationship
STOMATITIS (Gastrointestinal disorders) | 5 | 9 — Any Relationship
NAUSEA (Gastrointestinal disorders) | 4 | 13 — Any Relationship
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 | 0 — Any Relationship
CONSTIPATION (Gastrointestinal disorders) | 2 | 8 — Any Relationship
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 3 — Any Relationship
VOMITING (Gastrointestinal disorders) | 2 | 8 — Any Relationship
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 4 — Any Relationship
DRY MOUTH (Gastrointestinal disorders) | 1 | 2 — Any Relationship
DYSPEPSIA (Gastrointestinal disorders) | 1 | 5 — Any Relationship
FLATULENCE (Gastrointestinal disorders) | 1 | 2 — Any Relationship
GASTRITIS (Gastrointestinal disorders) | 1 | 1 — Any Relationship
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 | 0 — Any Relationship
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 | 0 — Any Relationship
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 — Any Relationship
MELAENA (Gastrointestinal disorders) | 0 | 2 — Any Relationship
ORAL DISORDER (Gastrointestinal disorders) | 0 | 2 — Any Relationship
ORAL PAIN (Gastrointestinal disorders) | 0 | 2 — Any Relationship
ASCITES (Gastrointestinal disorders) | 0 | 2 — Any Relationship
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 3 — Any Relationship
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0 — Any Relationship
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 6 — Any Relationship
FATIGUE (General disorders) | 7 | 22 — Any Relationship
CHEST DISCOMFORT (General disorders) | 2 | 1 — Any Relationship
CHILLS (General disorders) | 2 | 1 — Any Relationship
MUCOSAL INFLAMMATION (General disorders) | 2 | 5 — Any Relationship
OEDEMA PERIPHERAL (General disorders) | 2 | 12 — Any Relationship
PAIN (General disorders) | 2 | 2 — Any Relationship
CATHETER SITE PAIN (General disorders) | 1 | 0 — Any Relationship
DEATH (General disorders) | 1 | 0 — Any Relationship
DISEASE PROGRESSION (General disorders) | 1 | 0 — Any Relationship
EARLY SATIETY (General disorders) | 1 | 0 — Any Relationship
FACIAL PAIN (General disorders) | 1 | 0 — Any Relationship
OEDEMA (General disorders) | 1 | 0 — Any Relationship
PYREXIA (General disorders) | 1 | 4 — Any Relationship
ASTHENIA (General disorders) | 0 | 2 — Any Relationship
CHEST PAIN (General disorders) | 0 | 2 — Any Relationship
FACE OEDEMA (General disorders) | 0 | 2 — Any Relationship
ANAEMIA (Blood and lymphatic system disorders) | 5 | 9 — Any Relationship
NEUTROPENIA (Blood and lymphatic system disorders) | 5 | 12 — Any Relationship
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 3 — Any Relationship
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 3 — Any Relationship
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 2 — Any Relationship
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 2 — Any Relationship
URINARY TRACT INFECTION (Infections and infestations) | 3 | 7 — Any Relationship
HORDEOLUM (Infections and infestations) | 2 | 0 — Any Relationship
SINUSITIS (Infections and infestations) | 2 | 1 — Any Relationship
FUNGAL INFECTION (Infections and infestations) | 1 | 1 — Any Relationship
HERPES ZOSTER (Infections and infestations) | 1 | 0 — Any Relationship
NAIL INFECTION (Infections and infestations) | 1 | 0 — Any Relationship
ONYCHOMYCOSIS (Infections and infestations) | 1 | 0 — Any Relationship
PARONYCHIA (Infections and infestations) | 1 | 1 — Any Relationship
PNEUMONIA (Infections and infestations) | 1 | 2 — Any Relationship
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 8 — Any Relationship
URINARY TRACT INFECTION PSEUDOMONAL (Infections and infestations) | 1 | 0 — Any Relationship
VAGINAL INFECTION (Infections and infestations) | 1 | 0 — Any Relationship
CELLULITIS (Infections and infestations) | 0 | 2 — Any Relationship
INFECTION (Infections and infestations) | 0 | 2 — Any Relationship
RASH (Skin and subcutaneous tissue disorders) | 6 | 11 — Any Relationship
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 | 15 — Any Relationship
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 6 — Any Relationship
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 2 | 7 — Any Relationship
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 2 | 0 — Any Relationship
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 | 0 — Any Relationship
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 1 — Any Relationship
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 — Any Relationship
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 0 — Any Relationship
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 — Any Relationship
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1 | 0 — Any Relationship
ONYCHALGIA (Skin and subcutaneous tissue disorders) | 1 | 1 — Any Relationship
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 1 | 1 — Any Relationship
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 | 0 — Any Relationship
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 | 0 — Any Relationship
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 | 0 — Any Relationship
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 | 0 — Any Relationship
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 1 — Any Relationship
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 1 — Any Relationship
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 3 — Any Relationship
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 | 2 — Any Relationship
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 2 — Any Relationship
NEUROPATHY PERIPHERAL (Nervous system disorders) | 4 | 22 — Any Relationship
DYSGEUSIA (Nervous system disorders) | 3 | 2 — Any Relationship
DIZZINESS (Nervous system disorders) | 2 | 6 — Any Relationship
HEMICEPHALALGIA (Nervous system disorders) | 1 | 0 — Any Relationship
VISUAL FIELD DEFECT (Nervous system disorders) | 1 | 0 — Any Relationship
HEADACHE (Nervous system disorders) | 0 | 5 — Any Relationship
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 4 — Any Relationship
DYSARTHRIA (Nervous system disorders) | 0 | 3 — Any Relationship
HYPOAESTHESIA (Nervous system disorders) | 0 | 2 — Any Relationship
SCIATICA (Nervous system disorders) | 0 | 2 — Any Relationship
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 5 | 10 — Any Relationship
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 6 — Any Relationship
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 8 — Any Relationship
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — Any Relationship
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — Any Relationship
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Any Relationship
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 5 — Any Relationship
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Any Relationship
RHINORROEA (Respiratory, thoracic and mediastinal disorders) | 0 | 4 — Any Relationship
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 3 — Any Relationship
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 2 — Any Relationship
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 | 9 — Any Relationship
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 3 | 5 — Any Relationship
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 6 — Any Relationship
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 5 — Any Relationship
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 3 — Any Relationship
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 5 — Any Relationship
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 | 2 — Any Relationship
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 | 2 — Any Relationship
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 2 — Any Relationship
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 4 — Any Relationship
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 7 — Any Relationship
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 — Any Relationship
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 3 — Any Relationship
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 4 — Any Relationship
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 — Any Relationship
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 3 — Any Relationship
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 — Any Relationship
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 | 0 — Any Relationship
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 3 — Any Relationship
BACTERIAL TEST (Investigations) | 1 | 1 — Any Relationship
BLOOD CREATININE INCREASED (Investigations) | 1 | 1 — Any Relationship
HAEMATOCRIT DECREASED (Investigations) | 1 | 0 — Any Relationship
HEART RATE INCREASED (Investigations) | 1 | 0 — Any Relationship
SKIN TURGOR DECREASED (Investigations) | 1 | 0 — Any Relationship
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 | 1 — Any Relationship
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 | 0 — Any Relationship
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 5 — Any Relationship
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 | 4 — Any Relationship
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 3 — Any Relationship
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 3 — Any Relationship
WEIGHT DECREASED (Investigations) | 0 | 3 — Any Relationship
ANXIETY (Psychiatric disorders) | 2 | 2 — Any Relationship
DEPRESSION (Psychiatric disorders) | 2 | 2 — Any Relationship
INSOMNIA (Psychiatric disorders) | 2 | 5 — Any Relationship
DYSURIA (Renal and urinary disorders) | 2 | 5 — Any Relationship
NOCTURIA (Renal and urinary disorders) | 2 | 1 — Any Relationship
POLLAKIURIA (Renal and urinary disorders) | 1 | 0 — Any Relationship
URETHRITIS NONINFECTIVE (Renal and urinary disorders) | 1 | 0 — Any Relationship
URINARY TRACT PAIN (Renal and urinary disorders) | 1 | 0 — Any Relationship
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 2 | 1 — Any Relationship
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1 | 1 — Any Relationship
FALL (Injury, poisoning and procedural complications) | 1 | 0 — Any Relationship
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 — Any Relationship
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 2 — Any Relationship
EAR DISORDER (Ear and labyrinth disorders) | 1 | 0 — Any Relationship
VERTIGO (Ear and labyrinth disorders) | 1 | 0 — Any Relationship
CONJUNCTIVAL IRRITATION (Ear and labyrinth disorders) | 1 | 0 — Any Relationship
EYE PRURITUS (Ear and labyrinth disorders) | 1 | 0 — Any Relationship
OCULAR HYPERAEMIA (Ear and labyrinth disorders) | 1 | 0 — Any Relationship
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 1 | 0 — Any Relationship
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0 — Any Relationship
VULVOVAGINAL DISCOMFORT (Reproductive system and breast disorders) | 1 | 0 — Any Relationship
HOT FLUSH (Vascular disorders) | 1 | 2 — Any Relationship
LACRIMATION INCREASED (Eye disorders) | 0 | 3 — Any Relationship
CONJUNCTIVITIS (Eye disorders) | 0 | 2 — Any Relationship
VISION BLURRED (Eye disorders) | 1 | 2 — Any Relationship

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less